CLINICAL TRIAL: NCT06367881
Title: Assessment Of Dose-Dependent Immunomodulatory Effect Of Intratracheal Alveofact With Or Without Local Steroids In Respiratory Distress Syndrome Of Preterm Neonates
Brief Title: Assessment Of Dose-Dependent Immunomodulatory Effect Of Alveofact With or Without Steroisd In Neonatal RDS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amira Mostafa Rashad ibrahim, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD 185/ 2022
Record Dates: First submitted 2024-04-07; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Neonatal Respiratory Distress Syndrome; Inflammatory Response; Premature Lungs; Neutrophil Extracellular Trap Formation; Preterm Birth
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth | interventions — SF-RI 1, bovine surfactant preparation; Budesonide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Low dose Alveofact without steroids (Active Comparator): After obtaining parental consent, preterm neonates diagnosed with respiratory distress syndrome will be randomly administered a low dose of Intratracheal Alveofact (50 mg/kg) once without Budesonide. The clinical improvement of ventilatory settings, oxygen requirement, Assessment of Neutrophil Extracellular Trap (NET) formation, and Reactive Oxygen Species (ROS) will then be assessed before and 48 hours after treatment.
  The patient who will receive low-dose alveofact retreatment will be considered if the fraction of inspired oxygen (FiO2) was > 0.4 (does 50 mg/kg birth weight) 6 hours after treatment.
  Interventions: Drug: Alveofact
- Group 2: Low dose Alveofact with steroids (Experimental): After obtaining parental consent, preterm neonates diagnosed with respiratory distress syndrome will be randomly administered a low dose of Intratracheal Alveofact (50 mg/kg) once with Budesonide (0.25 mg/kg). The clinical improvement of ventilatory settings, oxygen requirement, Assessment of Neutrophil Extracellular Trap (NET) formation, and Reactive Oxygen Species (ROS) will then be assessed before and 48 hours after treatment.
  The patient who will receive low-dose alveofact retreatment will be considered if the fraction of inspired oxygen (FiO2) was > 0.4 (does 50 mg/kg birth weight) 6 hours after treatment.
  Interventions: Drug: Alveofact; Drug: Budesonide
- Group 3: High dose Alveofact without steroids (Active Comparator): After obtaining parental consent, preterm neonates diagnosed with respiratory distress syndrome will be randomly administered a High dose of Intratracheal Alveofact (100 mg/kg) once without Budesonide. The clinical improvement of ventilatory settings, oxygen requirement, Assessment of Neutrophil Extracellular Trap (NET) formation, and Reactive Oxygen Species (ROS) will then be assessed before and 48 hours after treatment.
  Interventions: Drug: Alveofact
- Group 4: Group 1: High dose Alveofact with steroids (Experimental): After obtaining parental consent, preterm neonates diagnosed with respiratory distress syndrome will be randomly administered a High dose of Intratracheal Alveofact (100 mg/kg) once with Budesonide(0.25 mg/kg). The clinical improvement of ventilatory settings, oxygen requirement, Assessment of Neutrophil Extracellular Trap (NET) formation, and Reactive Oxygen Species (ROS) will then be assessed before and 48 hours after treatment.
  Interventions: Drug: Alveofact; Drug: Budesonide

INTERVENTIONS:
Drug: Alveofact — Intratracheal High-dose Alveofact versus Low-dose Alveofact with or without Budesonide
Drug: Budesonide — Budesonide
  Arms: Group 2: Low dose Alveofact with steroids; Group 4: Group 1: High dose Alveofact with steroids

SUMMARY:
An Exploratory Randomized double-arm controlled trial to evaluate the immunomodulatory effect of low versus high dose of Alveofact with or without Budesonide.

DETAILED DESCRIPTION:
Neonatal respiratory distress syndrome (RDS) is caused by lung immaturity and surfactant deficiency in preterm newborns and is an important cause of morbidity and mortality.

Surfactant therapy plays an essential role in the management of RDS as it reduces lung injury and improves survival, While surfactant alone is very effective, some studies showed that its combination with budesonide significantly reduces BPD and inflammatory markers.

Neutrophils extracellular traps (NETs) are a defense mechanism where neutrophils are the reaction to microbial infection and cast a net-like structure. NETs are composed of chromatin decondensed and some 30 enzymes and peptides. Many components such as Neutrophil elastase (NE) and Myeloperoxidase enzyme (MPO) have antimicrobial, but also a cytotoxic property that causes tissue injury. The immune regulatory abilities of the pulmonary surfactant are known to alter the function of the adaptive and innate immune cells.

So, in this study, The Investigator will Assess the immunomodulatory effect of low and high doses of Alveofact with or without Budesonide.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≤ 35 weeks with

  1. Respiratory distress syndrome.
  2. Need surfactant administration based on European RDS consensus: (Sweet et al., 2019)
  3. If intubation is required as part of stabilization.
  4. Clinically presenting with increased work of breathing including (tachypnea, nasal flaring, grunting, retractions, and cyanosis, with decreased air entry on auscultation.
  5. Babies who are worsening when FiO2 >0.30 on CPAP pressure of at least 6 cm H2O to maintain normal saturations.

Exclusion Criteria:

Preterm neonates with evidence of any of the following will be excluded:

1. Chromosomal anomaly or Congenital heart defect
2. Hemodynamically significant patent ductus arteriosus.
3. Early-onset sepsis or bacterial infection
4. Congenital pneumonia
5. Intra ventricular hemorrhage (IVH)
6. Parenteral refusal to participate.

Ages: 1 Day to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of Neutrophil Extracellular Trap (NET) | 48 hours after treatment
  Neutrophil Extracellular Trapformation in neutrophil granulocytes as an evaluation of the therapeutic effect of two different doses of Alveofact with and without Steroids in Neonatal respiratory distress syndrome.
  Isolation of Neutrophil granulocytes from Bronchoalveolar fluid and whole blood samples using Neutrophil-specific magnetic beads. The purity and number of extracted neutrophils will be validated by cell morphology in hematoxylin-eosin staining and fluorescence-activated cell sorting for anti-CD-15 monoclonal antibodies.
  Assessment of Neutrophil Extracellular Trap (NET) formation: The amount of NET will be quantified by three different assays including; (1): measurement of neutrophil-specific Myeloperoxidase activity, (2): Neutrophil-elastase activity, and (3): Neutrophil-specific cell-free DNA (cfDNA).

SECONDARY OUTCOMES:
comparison of Alveolar with whole blood NET formation | 48 hours
  Neutrophil Extracellular Trap (NET) will be extracted in alveolar fluid and compared with whole blood samples
Clinical out come | 1 month
  Ventilation Duration in days.
Assessment of Reactive Oxygen Species (ROS) | 48 hours
  the lipid peroxidation will be calorimetrically measured using thiobarbituric acid (TBA) reactive compounds such as malondialdehyde (MDA) in microplates at 532 nm.
oxygen needs | 1 month
  FIO2 percentage on invasive and non-invasive respiratory support.
Hospital stay | 1 month
  Duration of NICU stay will be recorded in Days.

CONTACTS AND LOCATIONS:
Locations (1):
- Egypt Neonatal Intensive Care Units (NICUs), Ain Shams University Cairo, Abbasia, Egypt, 11517, Cairo, Egypt